CLINICAL TRIAL: NCT00812149
Title: Pharmacogenomic Response to Thyrotropin-Releasing Hormone Stimulation in Healthy Volunteers:The Influence of a Common Type 2 Deiodinase Genetic Polymorphism on Serum T3
Brief Title: Pharmacogenomic Response to Thyrotropin-Releasing Hormone Stimulation in Healthy Volunteers: The Influence of a Common Type 2 Deiodinase Genetic Polymorphism on Serum T3
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090058; 09-DK-0058
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2014-05-16

CONDITIONS: Thyroid Disease; Healthy
Keywords: Type-2 Deiodinase; Genetic Polymorphism; Triiodothyronine (T3); Thyrotropin Releasing Hormone (TRH) Test
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study intends to examine how a common genetic pattern affects thyroid function. Recent studies have demonstrated that a substance (enzyme) produced by a gene has an important role in controlling circulating thyroid hormone levels. A commonly found pattern in this gene exists in many individuals and might affect the function of the enzyme. These individuals need higher doses of thyroid hormone medication in certain situations (e.g. in the treatment of thyroid cancer after the thyroid gland has been removed) than those individuals without the variation.

We intend to study this by looking at the response to a hormone-test in healthy volunteers with different genetic patterns.

We plan to screen healthy volunteers using a blood test to identify their genetic pattern relating to the enzyme we are interested in. From this group, forty-five healthy volunteers will be recruited for the hormone-test. This test (called the TRH test) uses a hormone produced by the brain and stimulates the pituitary and thyroid gland. The response to this test will allow us to compare the function of the thyroid system in relation to the genetic pattern of the volunteer.

We hypothesize that the stimulation of the thyroid hormone system will be decreased in volunteers with a specific genetic pattern and that these individuals will release less active thyroid hormone from the thyroid gland in response to the TRH test.

This study will provide new information on the effect of a common genetic pattern on thyroid hormone function and will help us to better understand the way in which the thyroid hormone system operates. Ultimately, the results of this study might help to provide a more individualized therapy for patients in need of thyroid hormone replacement.

DETAILED DESCRIPTION:
This study intends to examine how a common genetic pattern affects thyroid function. Recent studies have demonstrated that a substance (enzyme) produced by a gene has an important role in controlling circulating thyroid hormone levels. A commonly found pattern in this gene exists in many individuals and might affect the function of the enzyme. These individuals need higher doses of thyroid hormone medication in certain situations (e.g. in the treatment of thyroid cancer after the thyroid gland has been removed) than those individuals without the variation.

We intend to study this by looking at the response to a hormone-test in healthy volunteers with different genetic patterns.

We plan to screen healthy volunteers using a blood test to identify their genetic pattern relating to the enzyme we are interested in. From this group, forty-five healthy volunteers will be recruited for the hormone-test. This test (called the TRH test) uses a hormone produced by the brain and stimulates the pituitary and thyroid gland. The response to this test will allow us to compare the function of the thyroid system in relation to the genetic pattern of the volunteer.

We hypothesize that the stimulation of the thyroid hormone system will be decreased in volunteers with a specific genetic pattern and that these individuals will release less active thyroid hormone from the thyroid gland in response to the TRH test.

This study will provide new information on the effect of a common genetic pattern on thyroid hormone function and will help us to better understand the way in which the thyroid hormone system operates. Ultimately, the results of this study might help to provide a more individualized therapy for patients in need of thyroid hormone replacement.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Subjects will be healthy male and female adult volunteers, between the ages of 18 and 65, able to provide informed consent. Patients younger than 18 are excluded as this is a purely physiologic study and we are unable to justify any potential risk. However, should our preliminary findings show potential clinically relevant benefits for children, the protocol could be modified to include them. Patients older than 65 are excluded due to intrinsic differences in thyroid hormone dynamics, compared with younger subjects, which could confound study interpretation.

EXCLUSION CRITERIA:

1. BMI less than or equal to 19 or greater than or equal to 35 Kg/m(2)
2. Hypothyroidism, or TSH levels above the normal limits (current replacement therapy or TSH greater than 4.0 mcIU/mL)
3. Hyperthyroidism, or TSH levels below the normal limits (current or previous therapy or TSH less than 0.4 mcIU/mL)
4. Autoimmune thyroid disease (as defined by a positive anti-TPO, or anti-TSH receptor antibody titer)
5. Hypertension (Blood pressure greater than 140/90 or use of antihypertensive medication)
6. Liver disease or ALT serum concentrations greater than 1.5 times the upper laboratory reference limit.
7. Renal insufficiency or estimated creatinine clearance less than or equal to 50 mL/min (MDRD equation).
8. History of, and/or current Diabetes Mellitus (fasting glucose greater than 126 mg/dL)
9. Iodine deficiency (spot urine iodine concentration less than 42 mcg/L)
10. History of, and/or current coronary artery disease
11. History of, and/or current asthma
12. History of, and/or current seizures or chronic headache
13. History of, and/or current depression
14. History of pituitary tumor
15. Pregnancy (women of child-bearing potential must have a negative pregnancy test prior to inclusion and at the time of TRH testing)
16. Known allergy to TRH
17. Current use of prescription medication or certain non-prescription medications and dietary supplements which could affect thyroid function and/or metabolism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-12-17; Study Completion 2014-05-16

CONTACTS AND LOCATIONS:
Overall Officials: Francesco S Celi, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bianco AC, Salvatore D, Gereben B, Berry MJ, Larsen PR. Biochemistry, cellular and molecular biology, and physiological roles of the iodothyronine selenodeiodinases. Endocr Rev. 2002 Feb;23(1):38-89. doi: 10.1210/edrv.23.1.0455. PMID 11844744
- [Background] Bianco AC, Kim BW. Deiodinases: implications of the local control of thyroid hormone action. J Clin Invest. 2006 Oct;116(10):2571-9. doi: 10.1172/JCI29812. PMID 17016550
- [Background] Bartha T, Kim SW, Salvatore D, Gereben B, Tu HM, Harney JW, Rudas P, Larsen PR. Characterization of the 5'-flanking and 5'-untranslated regions of the cyclic adenosine 3',5'-monophosphate-responsive human type 2 iodothyronine deiodinase gene. Endocrinology. 2000 Jan;141(1):229-37. doi: 10.1210/endo.141.1.7282. PMID 10614643
- [Derived] Butler PW, Smith SM, Linderman JD, Brychta RJ, Alberobello AT, Dubaz OM, Luzon JA, Skarulis MC, Cochran CS, Wesley RA, Pucino F, Celi FS. The Thr92Ala 5' type 2 deiodinase gene polymorphism is associated with a delayed triiodothyronine secretion in response to the thyrotropin-releasing hormone-stimulation test: a pharmacogenomic study. Thyroid. 2010 Dec;20(12):1407-12. doi: 10.1089/thy.2010.0244. Epub 2010 Nov 7. PMID 21054208